CLINICAL TRIAL: NCT06860503
Title: Clinical Characteristics and Thromboelastographic Evaluation of Hematotoxic Snakebites in Southern China: A 9-year Retrospective Study
Brief Title: Thrombelastography for Coagulopathy in Chinese Snakebites
Status: Completed | Type: Observational
Sponsor: Hansung University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20250218
Record Dates: First submitted 2025-02-18; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Pit Viper Bite; Coagulopathy; Thromboelastography (TEG); Venom-induced Consumptive Coagulopathy; Coagulation Disorder; Snake Envenomation; Disseminated Intravascular Coagulation (DIC)
Keywords: Pit Viper; TEG (Thromboelastography); Coagulopathy; Snake Bite; Venom-induced Coagulopathy; Clotting Disorders; Blood Coagulation Tests; Toxicology; Venomous Snake Bites
MeSH Terms: conditions — Hemostatic Disorders; Snake Bites; Disseminated Intravascular Coagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected from participants who have suffered pit viper bites. These samples will be used to perform coagulation tests, including thromboelastography (TEG) and traditional clotting tests (CCTs). The samples will be analyzed to assess coagulation disorders and the effectiveness of various diagnostic techniques. No DNA will be extracted or analyzed from these samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TEG group: Participants in this group are patients diagnosed with pit viper envenomation. They will undergo thromboelastography (TEG) testing to assess coagulation function. TEG testing will be performed at the time of hospital admission, as well as periodically during their treatment process, based on the clinical needs of each patient. The primary focus is on identifying coagulation abnormalities and monitoring changes over time.
- CCT group: Participants in this cohort are also diagnosed with pit viper envenomation, and they will undergo conventional coagulation tests (CCTs) such as PT, APTT, and fibrinogen levels. These tests will be used to monitor coagulation disorders and guide clinical management. The group will be compared to the TEG group to evaluate the effectiveness and accuracy of TEG in diagnosing venom-induced coagulopathy.

SUMMARY:
This study aims to evaluate the coagulation disorders caused by pit viper bites in patients from Zhanjiang and surrounding areas. The investigators will assess the effectiveness of thromboelastography (TEG) in evaluating coagulation function in these patients. The study will compare TEG results with conventional coagulation tests (CCTs) to understand its potential clinical value in diagnosing and managing coagulopathy caused by venomous snake bites.

DETAILED DESCRIPTION:
Pit viper bites are a significant cause of envenomation in Guangzhou and surrounding regions, leading to severe coagulation disorders. Early and accurate assessment of coagulation function is critical for effective management and treatment. Traditional coagulation tests, such as prothrombin time (PT) and activated partial thromboplastin time (APTT), are commonly used but may not fully reflect the complex coagulopathy induced by venom.

This observational study will include patients who have been bitten by pit vipers in Guangzhou and surrounding areas. The aim is to evaluate the role of thromboelastography (TEG) in the diagnosis and management of coagulopathy in these patients. The investigators will compare TEG results with conventional coagulation tests (CCTs) to assess their agreement and the additional insights TEG may provide in identifying coagulation abnormalities.

The study will observe participants from the moment of admission and monitor their coagulation function through TEG and CCTs. Data will be collected on clinical outcomes, including any signs of disseminated intravascular coagulation (DIC), thromboembolic events, or bleeding complications. The investigators aim to identify the clinical value of TEG in managing coagulopathy in pit viper bite cases and to explore whether TEG can be used as a more reliable and timely diagnostic tool.

This study will help improve the understanding of coagulopathy induced by pit viper venom and may potentially guide the development of better diagnostic and treatment protocols for venomous snake bites.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants aged 18-65 years.
* Diagnosis: Confirmed diagnosis of venom-induced consumptive coagulopathy caused by snake envenomation.
* Time of Enrollment: Participants who present with symptoms of venom poisoning within 6 hours of snake bite.
* Consent: Capable of providing written informed consent, or consent provided by a legal guardian if the participant is incapacitated.
* Vital Signs: Stable vital signs at the time of enrollment, with systolic blood pressure > 90 mmHg.
* Laboratory Results: Coagulation parameters (e.g., PT, aPTT, fibrinogen, platelet count) indicating acute coagulopathy.

Exclusion Criteria:

* Pregnancy or Breastfeeding: Women who are pregnant or breastfeeding.
* Severe Comorbidities: Participants with severe liver disease (e.g., cirrhosis), renal failure, or significant cardiovascular conditions (e.g., heart failure).
* Previous Snake Envenomation: Participants who have received antivenom for a snake bite in the past 30 days.
* Severe Allergies: Known allergy to snake venom antivenom or any of its components.
* Concurrent Participation in Other Clinical Trials: Participants who are currently enrolled in another clinical trial.
* Severe Coagulopathy or Bleeding Disorders: Participants with known pre-existing coagulation disorders such as hemophilia, or those with abnormal baseline blood tests suggesting coagulopathy unrelated to the snake bite.
* Immunocompromised Patients: Individuals with HIV/AIDS, or who are on immunosuppressive therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients aged 18 to 65 years diagnosed with venom-induced consumptive coagulopathy (VICC) following a pit viper snake bite. Participants must show clinical signs of envenomation (e.g., swelling, pain, coagulopathy such as prolonged PT, aPTT, low fibrinogen, and platelet count), confirmed by laboratory tests.
  Eligible patients will present to a medical facility within 6 hours of the bite and require antivenom treatment. Both male and female patients of all ethnicities will be included to reflect the general population affected by pit viper envenomation.
  Exclusion criteria include pregnancy, severe comorbidities, or known allergies to antivenom. Approximately 50 to 100 patients will be recruited to evaluate the clinical outcomes after antivenom treatment for VICC.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Thromboelastography (TEG) R (Reaction Time) in Pit Viper Bite Patients Thromboelastography (TEG) R (Reaction Time) in Pit Viper Bite Patients Thromboelastography (TEG) R (Reaction Time) in Pit Viper Bite Patients | Up to 24 hours
  This outcome measures the Reaction Time ® as part of the TEG assessment. R reflects the time to the initial clot formation and provides insight into the patient's ability to form a clot after a venomous pit viper bite. A prolonged R value may indicate a coagulation disorder.
Thromboelastography (TEG) K (Clot Formation Time) in Pit Viper Bite Patients | Up to 24 hours
  This outcome measures the Clot Formation Time (K) as part of the TEG analysis. K indicates the time it takes for the clot to form after the initial reaction, helping assess the speed of clot progression and the strength of coagulation. Prolonged K values may suggest fibrinogen deficiency or clotting factor depletion due to venom.
Thromboelastography (TEG) Alpha Angle in Pit Viper Bite Patients | Up to 24 hours
  This outcome measures the Alpha Angle, which reflects the rate of clot formation. A reduced Alpha Angle may indicate poor fibrinogen function or depletion, a key indicator of venom-induced coagulopathy.
Thromboelastography (TEG) Maximum Amplitude (MA) in Pit Viper Bite Patients | Up to 24 hours
  This outcome measures the Maximum Amplitude (MA), which assesses the strength of the clot. Decreased MA values could indicate weakened clot strength, a potential sign of venom-induced consumption coagulopathy. This helps identify patients at high risk of hemorrhagic complications.
Thromboelastography (TEG) Ly30 in Pit Viper Bite Patients | Up to 24 hours
  This outcome measures the Ly30, which represents the percentage of clot lysis 30 minutes after reaching maximum amplitude. Increased Ly30 values may indicate excessive fibrinolysis, which is common in patients with severe venom-induced coagulopathy.

SECONDARY OUTCOMES:
Mortality Rate | Up to 30 days
  This outcome measure assesses the mortality rate in patients with pit viper envenomation and venom-induced consumptive coagulopathy. Mortality is defined as death within 30 days following the bite.
Duration of Hospital Stay | From hospital admission to discharge
  This outcome measure evaluates the number of days patients remain in the hospital after being bitten by a pit viper and receiving antivenom treatment. The duration of stay is measured from the time of admission to discharge.
Incidence of Adverse Events | Up to 7 days
  This outcome measure tracks the occurrence of any adverse events related to antivenom administration or the progression of coagulopathy. Adverse events are categorized by severity (mild, moderate, severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Central People's Hospital of Zhanjiang, Zhanjiang, China